CLINICAL TRIAL: NCT02458612
Title: Effectiveness of Mirror Therapy Combined With Progressive Strength Training on Upper Limb Function in Children With Unilateral Spastic Cerebral Palsy
Brief Title: Effects of Mirror Therapy Combined With Progressive Strength Training in Unilateral Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, PT, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 15/135-43
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: cerebral palsy; mirror therapy; strength training
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): We will apply only upper limbs exercises with traditional therapy.
  Interventions: Other: control group
- intervention group (Active Comparator): We will apply mirror therapy and progressive strength training for upper extremities.
  Interventions: Other: intervention group

INTERVENTIONS:
Other: control group — We will apply traditional physiotherapy including upper limb exercises in three times a week for 12 week.
  Other Names: traditional therapy
  Arms: control group
Other: intervention group — Participants allocated to the experimental group completed three times a week, 12-week mirror therapy combined with progressive strength training. This protocol consisted of mirror therapy with a mirror box, strength training with Thera-band and exercises for scapular dyskinesis. This intensity of training is approximately equal to training at an intensity of 60% to 80% of one-repetition maximum according to "National Strength and Conditioning Association (NSCA)" protocols. Intensity of exercise is gradually increased 10% bi-weekly.
  Other Names: mirror therapy and progressive strength training
  Arms: intervention group

SUMMARY:
The purpose of this study is to investigate the effects of mirror therapy combined with upper extremity strengthening training on upper extremity function in children with unilateral spastic Cerebral Palsy (CP): a single blind randomized controlled trial. In the literature, there was no randomized controlled trial. According to literature, there are few studies that investigate the effects of mirror therapy in children with CP. But there is no randomized controlled trial, explore the effects of mirror therapy combined with upper extremity strength training on upper extremity functions in unilateral spastic CP. Hypothesis of this study is that mirror therapy combined with strength training improves upper extremity function and muscle strength in unilateral spastic CP.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a permanent but not progressive disorder of motor function and movement/posture that caused by lesion in the immature brain. Children with hemiplegic CP have unilateral motor disorder affecting the right or left half of the body. They constitute 42% of all CP. motor impairment of the upper extremity usually occurs more than the lower extremity. This motor impairment of upper extremity is one of the main reasons of the muscle weakness in children with unilateral CP. Nowadays studies has been proven to increase the activity and the body structure and function without any negative effect of strengthening education in children with CP. Park & Kim showed that huge impact of the upper and lower reinforcement training on children with CP the current meta-analysis (d = 0.861).

To improve upper extremity function in children with unilateral CP, the mirror therapy is a promising approach. Mirror therapy for the first time, Ramachandran et al. has described for the treatment of phantom pain in amputee. Also in unilateral spastic CP mirror therapy have indicated that visual illusion of functional limb provided by mirror can support healing. By means of visual feedback, modified vision and perception is stimulated plasticity the premotor cortex and developed reorganization. In the current studies, mirror therapy in hemiplegic patients, have been shown that improve the function and reduce the sensitivity of the hemi neglect. Gygax et al. have investigated the effects of mirror therapy on upper extremity function 10 children with unilateral spastic CP between 6-14 years. Consequently, the spontaneous use affected hand, the maximum grip force increase of 15% and is demonstrated that improve the upper extremity motor function.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 years and 18 years
* classified in levels I or II of the Gross Motor Function Classification System (GMFCS)
* classified in levels I, II-III of the Manual Ability Classification System (MACS)
* able to follow and accept verbal instructions.

Exclusion Criteria:

* any orthopaedic surgery or botulinum toxin injection in the past 6 months,
* children whose parents refused to participate
* Epileptic seizures that can not be stopped
* Individuals who can not participate in any physical activities because of chronic disease except cerebral palsy.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
upper extremity skills | change from baseline upper extremity skills at 12 weeks
  Quality of upper extremity skills assessment will be assessed by Quality of Upper Extremity Skills Test (QUEST). The test evaluates that handcraft and the quality of the movement in children with CP. It examines the quality of upper extremity skills in 5 sub-sections. It is used to between 18 monhts- 8 years age of children.

SECONDARY OUTCOMES:
muscle tone | change from baseline muscle tone at 12 weeks
  Children's muscle tone will be assessed by Modified Tardieu Scale (MTS). The original scale was developed in 1954 to assess spasticity by passive motion. This scale reveals the speed-dependent nature of spasticity. Passive stretching is made 3 different speeds that limb segment in the rate of fall with gravity and is faster than this speed and is slower than this speed. It has been developed by Boyd and Graham for 1999. Original scale is added to the assessment position of the limbs and angle of spasticity.
muscle strength | change from baseline muscle stregth at 12 weeks
  8 channels Biopac® MP150 surface electromyography for root mean square of maximum voluntary contraction, hand-held dynamometer "Power track II commander" for isometric muscle strength will be used to evaluate muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gygax MJ, Schneider P, Newman CJ. Mirror therapy in children with hemiplegia: a pilot study. Dev Med Child Neurol. 2011 May;53(5):473-6. doi: 10.1111/j.1469-8749.2011.03924.x. Epub 2011 Mar 17. PMID 21410693
- [Background] Piraua AL, Pitangui AC, Silva JP, Pereira dos Passos MH, Alves de Oliveira VM, Batista Lda S, Cappato de Araujo R. Electromyographic analysis of the serratus anterior and trapezius muscles during push-ups on stable and unstable bases in subjects with scapular dyskinesis. J Electromyogr Kinesiol. 2014 Oct;24(5):675-81. doi: 10.1016/j.jelekin.2014.05.009. Epub 2014 Jun 12. PMID 24997890
- [Background] Rameckers EA, Janssen-Potten YJ, Essers IM, Smeets RJ. Efficacy of upper limb strengthening in children with Cerebral Palsy: A critical review. Res Dev Disabil. 2015 Jan;36C:87-101. doi: 10.1016/j.ridd.2014.09.024. Epub 2014 Oct 15. PMID 25462469